CLINICAL TRIAL: NCT03316040
Title: Assessing the Impact of an Educational HIV Prevention Intervention in Zambia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: German Development Corporation (Other); American Institutes for Research (Other)
Responsible Party: Principal Investigator, Donald Green, Burgess Professor of Political Science, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAR2585
Record Dates: First submitted 2017-10-14; First posted 2017-10-20 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: HIV/AIDS
Keywords: HIV/AIDS; Join-in-Circuit
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Sex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control 1 (No Intervention): This arm represent control schools. No JIC will be implemented.
- Treatment 1 (Experimental): This arm implements the JIC among a random subset of students within the pre-defined grade.
  Interventions: Behavioral: JIC
- Treatment 2 (Experimental): This arm implements the JIC among indegree central students within the pre-defined grade.
  Interventions: Behavioral: JIC
- Treatment 3 (Experimental): This arm implements the JIC among edge betweeness central students within the pre-defined grade.
  Interventions: Behavioral: JIC

INTERVENTIONS:
Behavioral: JIC — The "Join In Circuit on HIV, love and sexuality" is a mobile learning system on the core topics of reproductive health and HIV and AIDS, targeting young people. JIC works with person-to-person communication in order to give an opportunity for discussion and for providing information in an open, engaging atmosphere. The JIC uses interactive exercises, pictorial aids and edutainment strategies to promote behavior change among young people aged 15 years and older.
  Other Names: Join-In-Circuit on AIDS, Love & Sexuality
  Arms: Treatment 1; Treatment 2; Treatment 3

SUMMARY:
In Zambia, 13% of the 15 to 49 year old population lives with HIV. The highest number of new HIV infections is among young people. To counter the spread of the disease, developmental and governmental actors are increasingly relying on educational behavior change tools. A particularly widely used tool, implemented by the German Development Corporation (henceforth, GIZ), is the so-called "Join-In-Circuit on AIDS, Love Sexuality" (JIC). The tool aims to improve a) HIV and sexual reproductive health knowledge, b) HIV testing uptake, and c) demand for health services. Previous research has investigated the direct effect of the JIC on knowledge about Sexually Transmitted Infections (STIs) as well as self-reported sexual behavior in Zimbabwe, and has found positive effects in both domains.

The research project evaluates the JIC in Zambia. The study randomly assigns 170 participating schools to five different JIC treatment arms. The first two arms represent control schools. Here, no JIC will be implemented. The third arm implements the JIC among a random subset of students. The fourth arm implements the JIC among indegree central students. The fifth arm implements the JIC among edge betweeness central students. In each school, the JIC will be implemented in one pre-determined grade. Within each school at least 30 students will be selected. For larger schools, 20 percent of students in the selected grade are selected.

DETAILED DESCRIPTION:
The study's population is schools in the Choma and Livingstone provinces of Zambia (a final set of 170 schools). The schools were provided by the Zambian Ministry of Education. The schools are split between primary (grade 1 to 7) and secondary schools (grade 8 to 12). In order to not interfere with exam periods, the Ministry of General Education and GIZ decided to implement the JIC among children in grade 6 in primary schools, and grade 11 in secondary schools.

On average, the schools have 80 students and 74 percent of the sample are in Choma. 88 percent of schools are considered rural, i.e., they do not lie in a major town. 4 percent of the sample have received a JIC before.

The 170 schools were randomly assigned to one of five treatment conditions.

* Control 1 (No intervention) (34 schools)
* Control 2 (No intervention) (34 schools)
* Treatment 1 (Random selection) (34 of schools)
* Treatment 2 (Indegree centrality) (34 of schools)
* Treatment 3 (Betweenness centrality) (34 of schools)

The Columbia University (CU) team advised GIZ on the design of the study, and the intervention will be solely run by GIZ. The CU team is not involved in the implementation of the study. Data will be collected by the American Institutes of Research (AIR). The CU team will only analyze fully de-identified data produced by the study.

ELIGIBILITY:
Inclusion Criteria:

* Students must be enrolled in the selected grade in one of the study schools and present on the day of the interview (for piloting) or on the day of baseline and endline (for main evaluation)
* Students must have informed consent
* Students must speak English or Tonga

Exclusion Criteria:

* There are no exclusion criteria within the pre-defined schools

Ages: 14 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 8270 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2017-12-02 (Actual); Study Completion 2017-12-02 (Actual)

PRIMARY OUTCOMES:
Standardized index of knowledge about sexual and reproductive health | Up to 6 months after the study implementation
  The investigators created an overall index that standardizes the outcome variables, which is split into a knowledge index and a self-reported behavior. This index will be constructed from a battery of survey items pertaining to knowledge about condoms, HIV/Aids and other STIs.

SECONDARY OUTCOMES:
Standardized index of self-reported behavior | Up to 6 months after the study implementation
  The investigators created an overall index that standardizes the outcome variables, which is split into a knowledge index and a self-reported behavior. This index will be constructed form a battery of survey items measuring self-reported behavior pertaining to sex, HIV testing, and access of health facilities.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Green, PhD, Principal Investigator — Columbia University
Locations (3):
- Columbia University, New York, New York, United States
- Zambia (2):
  - American Institutes for Research, Choma
  - American Institutes for Research, Livingstone

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Statistical Analysis Plan (2017-10-13): https://cdn.clinicaltrials.gov/large-docs/40/NCT03316040/SAP_001.pdf